CLINICAL TRIAL: NCT06742892
Title: A Phase II Clinical Study to Evaluate HLX43 (Anti-PD-L1 ADC) in Patients With Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC) Failed or Intolerance to Standard Therapy
Brief Title: A Phase II Clinical Study to Evaluate HLX43 in Patients With Locally Advanced or Metastatic HCC Failed or Intolerance to Standard Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX43-HCC201
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLX43 DOSE 1 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 1
- HLX43 DOSE 2 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 2
- HLX43 DOSE 3 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 DOSE 3

INTERVENTIONS:
Drug: HLX43 DOSE 1 — Dose 1; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Anti-PD-L1 ADC
  Arms: HLX43 DOSE 1
Drug: HLX43 DOSE 2 — Dose 2; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Anti-PD-L1 ADC
  Arms: HLX43 DOSE 2
Drug: HLX43 DOSE 3 — Dose 3; HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Other Names: Anti-PD-L1 ADC
  Arms: HLX43 DOSE 3

SUMMARY:
The study is being conducted to to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC) Failed or Intolerance to Standard Therapy

DETAILED DESCRIPTION:
This study is an open-label phase II clinical study to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in Patients with Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC) Failed or Intolerance to Standard Therapy. In this study, eligible subjects will be randomized at 1:1:1 ratio, and the patients will be administered with HLX43 at different doses via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research;To fully understand and understand this study and to sign the Informed Consent Form (ICF);Willing to follow and able to complete all test procedures
2. The age of signing ICF is ≥ 18 years old and ≤ 75 years old，regardless of gender;
3. Hepatocellular carcinoma (HCC) confirmed by histopathology or cytology, or clinically meeting the American Association of Hepatology (AASLD) criteria for HCC diagnosis；
4. Previous failure or progression of at least one standard systemic therapy for hepatocellular carcinoma (standard therapy refers to PD-1/ L1-based combination therapy, or lenvatinib, sorafenib), or intolerability toxicity (CTCAE≥3 adverse events), or contraindications to standard therapy.
5. Barcelona Clinic Liver Cancer (BCLC) stage C; BCLC stage B patients who are not suitable for locoregional therapy may also be enrolled.
6. Within 4 weeks prior to the first administration of the medication, at least one measurable target lesion must be evaluated according to the RECIST v1.1 criteria. A region that has received prior local treatment may also be selected as a target lesion if there is a clear progression that meets the RECIST v1.1 standards；
7. Tumor tissue should be provided as much as possible for an evaluable PD-L1 expression result at Screening period；
8. Before the initial administration of the study drug, there should be at least a 3-week interval or 5 times the half-life of the last cytotoxic chemotherapy, immunotherapy, or biological therapy, whichever is shorter. There should be at least a 2-week interval from the previous small molecule targeted therapy, at least a 1-week interval from traditional Chinese medicine treatment with antitumor indications or minor surgery. Additionally, treatment-related adverse events (AEs) should have recovered to NCI-CTCAE grade ≤ 1 (except for grade 2 peripheral neurotoxicity and alopecia)；
9. Child-pugh liver function rating within 7 days before the first administration of the study drug : grade A；
10. The ECOG physical performance score of 0-1 in the week prior to randomization；
11. Expected survival ≥ 3 monthes；
12. Subjects of HBsAg (-) and HBcAb (-) are allowed to be enrolled. If HBsAg (+) or HBcAb (+), then HBV-DNA must be < 500 IU/mL or <2500 copy/ml or <ULN to be eligible for enrollment. Subjects with negative HCV antibodies (-) or negative HCV-RNA are allowed to be included in the study. Subjects with negative HCV antibodies (-) or negative HCV-RNA are allowed to be included in the study. If HCV-RNA is positive, consent must be obtained to receive the local standard antiviral treatment, and participants must have ALT and AST levels ≤ 3×ULN to be eligible for enrollment. Subjects with co-infection of hepatitis B and hepatitis C need to be excluded (both HBV-DNA and HCV-RNA are positive)；
13. Laboratory tests within the previous week confirm adequate organ function (within 14 days prior to the first dose of medication, without receiving interventions such as blood transfusions or granulocyte colony-stimulating factor)；
14. Male and female subjects of childbearing potential must agree to use at least one highly effective method of contraception during the trial and for at least 6 months after the last dose of the study drug. Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

1. Hepatobiliary duct cell carcinoma, mixed cell carcinoma, or fibroblastic layer cell carcinoma are known;
2. History of any second malignant tumor within the first 2 years prior to randomization, excluding early-stage malignancies that have been treated curatively (carcinoma in situ or stage I tumors), such as non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, breast ductal carcinoma in situ, and papillary thyroid carcinoma;
3. History of hepatic encephalopathy or has undergone a liver transplant. Patients who are preparing for or have previously undergone organ or bone marrow transplantation;
4. Within 6 months prior to randomization, present with portal hypertension accompanied by upper gastrointestinal bleeding, or have esophageal/gastric varices with red wale markings, or are at risk of ruptured hemorrhagic hepatic cancer nodules, or are considered by the researcher to be at high risk of bleeding;
5. According to the images, portal vein invasion, inferior vena cava or cardiac involvement of HCC main portal branch (Vp4) were present. Patients with cancer thrombus in main portal vein but smooth blood flow in contralateral branch can be enrolled;
6. After appropriate intervention, uncontrollable pleural effusion, pericardial effusion or ascites still need to be drained frequently;
7. Symptomatic, untreated, or progressively worsening central nervous system (CNS) or leptomeninges metastases;
8. Received major surgery or any local treatment targeting liver lesions (including but not limited to surgery, radiotherapy, hepatic artery embolization, transcatheter arterial chemoembolization (TACE), hepatic artery infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection) within 4 weeks prior to randomization;
9. Received radiation therapy within the last 4 weeks and abdominal/pelvic radiation therapy within the previous 8 weeks, excluding palliative radiation therapy for bone disease;
10. Patients with previous and current cases of interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, and severe impairment of lung function that may interfere with the detection and management of suspected drug-related lung toxicity;
11. Known history of severe allergic reactions to macromolecular protein preparations/monoclonal antibodies, or allergy to components of the trial drug formulation;
12. Within the 2 weeks prior to randomization, there is the presence of an active systemic infectious disease requiring intravenous antibiotic treatment;
13. Subjects exhibit poorly controlled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or above heart failure, or left ventricular ejection fraction (LVEF) < 50%; (2) unstable angina; (3) myocardial infarction or cerebrovascular accident within the last 6 months (excluding lacunar infarction, minor ischemic stroke, or transient ischemic attack); (4) uncontrolled arrhythmias (including QTc interval ≥ 450 ms for males, ≥ 470 ms for females) (QTc interval calculated by Fridericia's formula); (5) poorly controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg despite active treatment);
14. A history of ≥ Grade 3 immune-related adverse events during previous immunotherapy;
15. Active or suspected autoimmune disease. Patients with autoimmune-related hypothyroidism who are undergoing thyroid hormone replacement therapy are permitted to participate in the study; patients with controlled Type 1 diabetes mellitus receiving insulin therapy are also allowed to participate in the study;
16. Received systemic corticosteroids (prednisone >10 mg/day or an equivalent dose of similar drugs) or other immunosuppressive treatments within 14 days prior to the first dose; with the following exceptions: use of topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids; short-term use of corticosteroids for prophylactic treatment during situations such as the use of contrast agents;
17. Live vaccinations or attenuated live vaccinations should not be administered within 4 weeks prior to the initial dosing. Administration of inactivated viral vaccines for seasonal influenza is permitted;
18. Used strong inhibitors or strong inducers of CYP2D6 or CYP3A within 2 weeks prior to randomization;
19. Active tuberculosis
20. Human immunodeficiency virus (HIV) infection;
21. Pregnant or lactating women;
22. The researcher deems that the subject has any other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 week
  Objective response rate (ORR) (assessed by INV according to the RECIST v1.1 criteria)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV according to the RECIST v1.1 criteria.

SECONDARY OUTCOMES:
ORR | up to 24 weeks
  Objective response rate (ORR) (assessed by the IRRC according to the RECIST v1.1 criteria)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 14 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC according to the RECIST v1.1 criteria.
OS | From randomization to death from any cause (up to approximately 36 months)
  Overall Survival
Incidence and severity of adverse events (AEs) | time from the date of the first dose of study drug until the date of death from any cause, assessed up to 24 months
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0, vital signs and clinical laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Hua Xiang, Dr., Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Hunan, Hunan, China